CLINICAL TRIAL: NCT02641574
Title: Relation Between Complication in Repeated Cesarean Sections Compared With Newborn Outcome,Surgical Characteristics and Maternal Information
Brief Title: Relation Between Complication in Repeated Cesarean Sections, Newborn Outcome and Surgical Characteristics and Maternal Information
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yechiel Burke MD, Doctor, Rambam Health Care Campus
Other Study IDs: 102892
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Women Who Had at Lease One Cesarean Section in the Past

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (4):
- previous 1: women who have had in their past one cesarean section
  Interventions: Other: compare complication
- previous 2: women who have had in their past 2 cesarean sections
  Interventions: Other: compare complication
- previous 3: women who have had in their past 3 cesarean sections
  Interventions: Other: compare complication
- previous 4: women who have had in their past 4 cesarean sections
  Interventions: Other: compare complication

INTERVENTIONS:
Other: compare complication

SUMMARY:
To examine the relation between complication in Repeated Cesarean Sections and Newborn Outcome compared to number of repeated cesarean section and reasonf or surgery and personal medical information to the mother

ELIGIBILITY:
Inclusion Criteria:

women who had at least one cesarean section -

Exclusion Criteria:

women that this was their first cesarean section

-

Ages: 17 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All women who underwent a cesarean section at Rambam Medical Center who had at least one cesarean section in the past
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2009-01; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
surgical complication compared to number of repeated cesarean sections | during the surgery